CLINICAL TRIAL: NCT03350659
Title: Efficacy and Safety of Midodrine and Atomoxetine Treatment in Patients With Neurogenic Orthostatic Hypotension : A Prospective Randomized Study
Brief Title: Efficacy and Safety of Midodrine and Atomoxetine for Neurogenic OH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, Kon Chu, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1710-060-893
Record Dates: First submitted 2017-11-18; First posted 2017-11-22 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Neurogenic Orthostatic Hypotension
Keywords: orthostatic hypotension; midodrine; atomoxetine; treatment
MeSH Terms: conditions — Hypotension, Orthostatic | interventions — Midodrine; Atomoxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Randomized, open-label clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atomoxetine (Experimental): Atomoxetine 18mg once a day.
  Interventions: Drug: Atomoxetine
- Midodrine (Active Comparator): midodrine 2.5mg twice a day (increase to 5mg three times a day if necessary)
  Interventions: Drug: Midodrine

INTERVENTIONS:
Drug: Midodrine — Midodrine single 5mg/day
  Other Names: Midodrine only
  Arms: Midodrine
Drug: Atomoxetine — Atomoxetine single 18mg/day
  Other Names: Atomoxetine only
  Arms: Atomoxetine

SUMMARY:
This was a randomized, open-label clinical trial. We will enroll patients with symptomatic neurogenic OH and randomize them to 1 of 2 treatments: (1) midodrine only, (2) atomoxetine only. We will follow up patients at 1 and 3 months after treatment. If the patients meet BP criteria for OH at 1 month, they will receive combination treatment with both midodrine and atomoxetin. The primary outcome measure is amelioration of questionnaire score evaluating OH-associated symptoms at 3 months. Secondary end-points were improvement in orthostatic blood pressure (BP) drop at 1 and 3 months.

DETAILED DESCRIPTION:
Visit 1.

1. Enroll, baseline evaluation of the patients
2. Questionnaire

   * Evaluate orthostatic hypotension symptom: Orthostatic Hypotension Questionnaire (OHQ)
   * Quality of life: Korean version of Short-form 36
   * Depressive symptom: Korean version of Beck Depression Inventory(BDI)-2
3. Blood test (6cc): ELISA for alpha 1,2 and beta 1,2 adrenergic receptor antibody and nicotinic acetylcholine receptor antibody. Preserve sample for genetic testing.
4. Randomization: randomize patients to three group in 1:1 ratio (Midodrine 5mg/day single, Atomoxetine 18mg/day single)
5. Treatment education Visit 2. 1 month after treatment Orthostatic BP check/ check drug compliance and side effect/ Questionnaire If the patients meet BP criteria for OH, initiate combination treatment (Midodrine 5mg/day+Atomoxetine 18mg/day) Visit 3. 3 months after treatment Orthostatic BP check/ check drug compliance and side effect/ Questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Age >=19 patients who complained of dizziness
* Orthostatic hypotension after 3-minute standing (systolic blood pressure drop >=20 or diastolic blood pressure drop >=10

Exclusion Criteria:

* Drug-induced hypotension, if necessary, evaluate patient after discontinuing the causative drug for one month
* Heart failure or Chronic renal failure
* Severe supine hypertension (Systolic Blood Pressure >180 or Diastolic Blood Pressure>110mmHg)
* Pregnant women, breast-feeding
* Unable to perform questionnaire

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Change of the Orthostatic Hypotension Associated Symptom Questionnaire (OH Questionnaire (OHQ) | after 3-month medical treatment
  Change of the OH associated symptom survey result after 3-month medical treatment compared to initial results. OHQ questionnaire has two components: the OH daily activity scale (OHDAS), which contains 4 items measuring the impact of OH on daily activities, and the OH symptom assessment (OHSA), which contains 6 items measuring the symptoms of OH (dizziness/light headedness, vision disturbance, weakness, fatigue, trouble concentrating, and head/neck discomfort).This questionnaire reflects the severity of OH-related symptoms on a 10-point scale, with 0 indicating the absence of a symptom and 10 indicating maximal severity.
  ** OHQ total score minimal 0 ~ maximal 100 (subscale OHDAS score minimal 0~ maximal 40, OHSA score minimal 0~ maximal 60)

SECONDARY OUTCOMES:
Change in Orthostatic blood pressure Drop (mmHg) | after 3-month medical treatment
  Change of orthostatic Systolic blood pressure and Diastolic Blood Pressure drop after 3-month medical treatment compared to initial results.
Change of the Depression Score (Beck Depression Inventory-II ) | after 3-month medical treatment
  Change of the depression score after 3-month medical treatment compared to initial results.
  21 multiple-choice questions, each of which can be scored from 0 to 3. Higher score represent higher degree of depression. Score Normal; 0-13, Mild depression; 14-19, Moderate depression; 20-28, Severe depression; 29- 63
Changes in Health-related Quality of Life | after 3-month medical treatment
  changes in Short Form (36) Health Survey version 2 (SF-36v2) physical component summary scale (PCS) compared to the baseline SF-36v2 measures eight HRQOL domains (physical functioning, role limitation caused by physical problems, bodily pain, general health, vitality, social functioning, role limitation caused by emotional problems, and mental health) summarized into two summary scales that are normalized to the population (mean=50, standard deviation=10): the physical component summary scale (PCS) and the mental component summary scale (MCS).20 Better HRQOL is reflected by higher SF-36v2 scores.

CONTACTS AND LOCATIONS:
Overall Officials: Chu Kon, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Consensus statement on the definition of orthostatic hypotension, pure autonomic failure, and multiple system atrophy. The Consensus Committee of the American Autonomic Society and the American Academy of Neurology. Neurology. 1996 May;46(5):1470. doi: 10.1212/wnl.46.5.1470. No abstract available. PMID 8628505
- [Background] Smit AA, Halliwill JR, Low PA, Wieling W. Pathophysiological basis of orthostatic hypotension in autonomic failure. J Physiol. 1999 Aug 15;519 Pt 1(Pt 1):1-10. doi: 10.1111/j.1469-7793.1999.0001o.x. PMID 10432334
- [Background] Hiitola P, Enlund H, Kettunen R, Sulkava R, Hartikainen S. Postural changes in blood pressure and the prevalence of orthostatic hypotension among home-dwelling elderly aged 75 years or older. J Hum Hypertens. 2009 Jan;23(1):33-9. doi: 10.1038/jhh.2008.81. Epub 2008 Jul 24. PMID 18650837
- [Background] Hale GM, Valdes J, Brenner M. The Treatment of Primary Orthostatic Hypotension. Ann Pharmacother. 2017 May;51(5):417-428. doi: 10.1177/1060028016689264. Epub 2017 Jan 16. PMID 28092986
- [Background] Low PA, Singer W. Management of neurogenic orthostatic hypotension: an update. Lancet Neurol. 2008 May;7(5):451-8. doi: 10.1016/S1474-4422(08)70088-7. PMID 18420158
- [Background] Wright RA, Kaufmann HC, Perera R, Opfer-Gehrking TL, McElligott MA, Sheng KN, Low PA. A double-blind, dose-response study of midodrine in neurogenic orthostatic hypotension. Neurology. 1998 Jul;51(1):120-4. doi: 10.1212/wnl.51.1.120. PMID 9674789
- [Background] Parsaik AK, Singh B, Altayar O, Mascarenhas SS, Singh SK, Erwin PJ, Murad MH. Midodrine for orthostatic hypotension: a systematic review and meta-analysis of clinical trials. J Gen Intern Med. 2013 Nov;28(11):1496-503. doi: 10.1007/s11606-013-2520-3. Epub 2013 Jun 18. PMID 23775146
- [Background] Izcovich A, Gonzalez Malla C, Manzotti M, Catalano HN, Guyatt G. Midodrine for orthostatic hypotension and recurrent reflex syncope: A systematic review. Neurology. 2014 Sep 23;83(13):1170-7. doi: 10.1212/WNL.0000000000000815. Epub 2014 Aug 22. PMID 25150287
- [Background] Byun JI, Moon J, Kim DY, Shin H, Sunwoo JS, Lim JA, Kim TJ, Lee WJ, Lee HS, Jun JS, Park KI, Lee ST, Jung KH, Jung KY, Lee SK, Chu K. Efficacy of single or combined midodrine and pyridostigmine in orthostatic hypotension. Neurology. 2017 Sep 5;89(10):1078-1086. doi: 10.1212/WNL.0000000000004340. Epub 2017 Aug 9. PMID 28794253
- [Background] Ramirez CE, Okamoto LE, Arnold AC, Gamboa A, Diedrich A, Choi L, Raj SR, Robertson D, Biaggioni I, Shibao CA. Efficacy of atomoxetine versus midodrine for the treatment of orthostatic hypotension in autonomic failure. Hypertension. 2014 Dec;64(6):1235-40. doi: 10.1161/HYPERTENSIONAHA.114.04225. Epub 2014 Sep 2. PMID 25185131
- [Background] Hale GM, Brenner M. Atomoxetine for Orthostatic Hypotension in an Elderly Patient Over 10 Weeks: A Case Report. Pharmacotherapy. 2015 Sep;35(9):e141-8. doi: 10.1002/phar.1635. PMID 26406777